CLINICAL TRIAL: NCT00145873
Title: Continuous Infusion Nesiritide in Chronic Heart Failure-University of Chicago (CINCH-UC)
Brief Title: Nesiritide in Chronic Heart Failure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to complete study
Sponsor: University of Chicago (Other)
Collaborators: Scios, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 12350A; 1
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2006-09

CONDITIONS: Heart Failure
Keywords: heart failure; nesiritide; heart disease; cardiovascular disease
MeSH Terms: conditions — Heart Failure; Heart Diseases; Cardiovascular Diseases | interventions — Natriuretic Peptide, Brain

INTERVENTIONS:
Drug: nesiritide, continuous infusion

SUMMARY:
The purpose of this study is to look at the safety and effectiveness of longer term intravenous (IV) infusion of the study drug, nesiritide in patients with acutely decompensated chronic heart failure. Nesiritide (Natrecor) is a man-made version of a human hormone that dilates veins and arteries. Nesiritide (Natrecor) is currently FDA-approved for short-term inpatient IV treatment of acutely decompensated chronic heart failure.

Hypothesis: Nesiritide, administered by continuous intravenous infusion in the outpatient setting, is a safe treatment for refractory Class III & IV chronic heart failure due to systolic or diastolic dysfunction, regardless of renal function when administered over a 12-week period.

Corollary #1: Nesiritide, when infused continuously over 12 weeks will improve the overall condition of patients with chronic heart failure. These mechanisms include reducing hospitalizations when compared with the previous six months, improving symptoms as measured by the Minnesota Living with Heart Failure short questionnaire, and improving functional capacity as measured by 6-minute walk testing.

Corollary #2: Nesiritide infusion will be associated with a statistically significant decrease in N-terminal pro-BNP levels and cyclic GMP levels compared with patients receiving placebo infusions.

DETAILED DESCRIPTION:
This is a single center, double-blinded, crossover, placebo-controlled pilot study to evaluate the effects of nesiritide in patients with chronic heart failure. This study will only take place at the University of Chicago Hospitals. It is double-blinded, which means that the neither subject nor their study doctor will know which study drug the subject will receive. However, in an emergency, this information can be obtained quickly. The study is placebo-controlled, which means subjects will not receive study drug at some point during the study; however because it is a cross-over study, subjects will be receiving nesiritide at some point in the study. Subjects will receive the study drug nesiritide for six out of the 12 weeks of the study-either the first six weeks or the last six weeks.

The procedures for the study consist of: informed consent, questions about the subjects heart failure, blood sample, assessment of heart failure severity based on symptoms, six minute walk test and the Minnesota Living with Heart Failure Questionnaire, history of heart failure symptoms and emergency room visits, diuretic and baseline medication history, long term IV for medication infusions, adjustment of study drug and regularly taken medications, 6 weeks of receiving long term IV infusion of drug, blood taken for lab tests at each clinic visit and an informational card provided for subjects to use for on-call physicians.

Up to ten consecutive patients who decline participation in the study will be asked to participate in a registry to follow their course over the study interval. Baseline data, obtained from medical records will be recorded as will the number of hospitalizations/ER visits and NYHA class during the study period. These subjects will be surveyed by telephone monthly for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

Candidates for enrollment in this clinical trial are limited to adult patients (age>21) diagnosed with chronic heart failure > one year who are managed by heart failure specialists at the University of Chicago. Patients primarily managed by physicians other than the investigators will be enrolled with the concurrence of the treating physician. Study patients are characterized as "high risk" by fulfilling one or more of the following criteria:

1. Refractory class III or IV heart failure despite optimal medical therapy by a heart failure specialist: Angiotensin converting enzyme inhibitors (ACEI), angiotensin receptor blockers (ARB), beta-adrenergic blockers (BB), spironolactone (spiro), digoxin (dig), diuretics, and calcium channel blockers (CCB).
2. Frequent hospitalizations or ER visits (>1/month on average).

Additionally, patients must be capable of giving informed consent and have adequate social supports to manage chronic, continuous IV infusion therapy with the assistance of home care nursing and the study coordinator.

Exclusion Criteria:

1. Nesiritide infusion >24 hours in the previous 30 days.
2. Stable chronic heart failure or NYHA Class I or II.
3. Aortic stenosis greater than mild degree as determined by echocardiogram or catheterization.
4. Hypertrophic cardiomyopathy with an outflow tract gradient.
5. Isolated right heart failure (cor pulmonale).
6. Unstable coronary syndrome or myocardial infarction< 3 months prior to enrollment.
7. Chronic hypotension with systolic blood pressure < 80 mmHg.
8. Terminal noncardiovascular illness with life expectancy <6 months. Moribund patients will not be considered for enrollment.
9. Active substance abuse.
10. Inadequate social support.
11. Contraindication to long term IV access.
12. Pregnant or lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2003-08; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Change in NYHA status | Day 0, Day 42

CONTACTS AND LOCATIONS:
Overall Officials: Allen Anderson, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Hospitals, Chicago, Illinois, United States